CLINICAL TRIAL: NCT01142089
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Rifamycin SV MMX for the Treatment of Traveler's Diarrhea
Brief Title: Study to Evaluate Safety and Efficacy of Rifamycin SV Multi-Matrix System (MMX) for the Treatment of Traveler's Diarrhea (TD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2009-0201
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-04

CONDITIONS: Traveler's Diarrhea
Keywords: traveler's; diarrhea; Rifamycin SV MMX; Rifamycin; MMX; Traveler's Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (two matching tablets) orally twice daily for 3 days (72 hours)
  Interventions: Drug: Placebo
- Rifamycin SV MMX (Experimental): Rifamycin SV MMX® 400 mg (two 200 mg tablets) orally twice daily for 3 days (72 hours).
  Interventions: Drug: Rifamycin SV MMX

INTERVENTIONS:
Drug: Placebo — Placebo (two matching tablets) orally twice daily for 3 days (72 hours).
  Arms: Placebo
Drug: Rifamycin SV MMX — Rifamycin SV MMX® 400 mg (two 200 mg tablets) orally twice daily for 3 days (72 hours).
  Arms: Rifamycin SV MMX

SUMMARY:
The purpose of this study is to determine whether Rifamycin SV MMX is a safe and effective treatment for Traveler's Diarrhea.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled efficacy and safety study conducted in patients traveling to developing regions with a known high incidence of TD. Eligibility will be based on a symptom complex that is highly indicative of enteric acute bacterial infection without indication of systemic infection.

Approximately 262 patients will be enrolled in the study and randomized at a 3:1 ratio to receive Rifamycin SV MMX® 400 mg or placebo orally twice daily for 3 days (72 hours). Treatment will be initiated on the day of Screening (Visit 1, Day 1), within 72 hours of onset of diarrhea. Daily doses of study drug will be taken at breakfast time and dinner time with a glass of liquid.

Safety and efficacy will be assessed.

Blood samples for routine safety tests (chemistry and hematology) will be collected at Visit 1 and at Visit 3 and sent to a local laboratory for analysis and reporting to the Investigator for safety monitoring. Urine samples for routine urinalysis (dipstick only) will be collected at Visits 1 and 3, and the results will be used by the Investigator for safety monitoring.

If a patient's diarrhea and/or signs or symptoms of enteric infection worsen in a 24 hour interval of time during the treatment period or if the enteric illness fails to improve after 24 hours or more of therapy, the patient may receive Rescue Therapy. Rescue Therapy will be prescribed by the Investigator using local standard empiric therapy and/or guided by pathogen identification.

ELIGIBILITY:
Inclusion Criteria

Patients were enrolled in the study only if they met all of the following criteria:

1. Male and female patients 18 years of age or older
2. Female and male patients of childbearing potential must have agreed to use an effective method of birth control (this method must have been approved by the investigator and may have included total abstinence from sexual intercourse) during the treatment and follow-up study periods; female patients of childbearing potential must have had a negative pregnancy test in the 72 hours before randomization; female patients who abstained totally from sexual intercourse were not required to take the pregnancy test
3. Recent travel (i.e., must be within 30 days of randomization) from an industrialized country
4. Experiencing signs or symptoms indicative of acute bacterial diarrhea (TD), defined as at least three unformed, watery or soft, stools within the 24 hours preceding randomization and the duration of illness 72 hours before randomization, and able to provide an unformed stool sample during Screening (the latter can be the third unformed stool passed by the patient within the 24 hours preceding randomization); the bacterial cause of diarrhea was confirmed by microbiology analysis of the stool sample
5. Experiencing one or more signs or symptoms of enteric infection (moderate to severe gas/flatulence, nausea, vomiting, abdominal cramps or pain, rectal tenesmus, or defecation urgency)
6. Capable of and willing to give informed consent

Exclusion Criteria

Patients were excluded from the study if they met any of the following criteria:

1. Fever (> 100.4F or 38C) or presence of signs and symptoms of systemic infection Note: antipyretic medication should not have been administered in the 6 hours before this assessment
2. Known or suspected infection with non-bacterial pathogen before randomization
3. Presence of diarrhea for > 72 hours duration
4. Presence of grossly bloody stool
5. Presence of moderate to severe dehydration (i.e., presence of orthostatic hypotension and/or dehydration requiring treatment with intravenous fluids)
6. History of ulcerative colitis, diarrhea-predominant irritable bowel syndrome, Crohn's disease, celiac sprue (gluten-enteropathy), chronic pancreatitis, malabsorption, or any other gastrointestinal disease associated with diarrhea. Note: lactose intolerance treated with lactase supplements or a lactose-free diet were not excluded if these regimens were maintained during the study.
7. Receiving more than two doses of an antidiarrheal medication (e.g., antimotility, absorbent, adsorbent, antisecretory, or probiotics) within 24 hours before randomization
8. Receiving one or more of the following antibiotics, which are active against gram negative bacteria TMP-SMX, fluorquinolone, azithromycin or rifaximin within 7 days before randomization
9. Females pregnant or breast feeding or not using adequate birth control
10. Known intolerance/hypersensitivity/resistance to rifamycin or rifamycin-related antibiotics or to any excipient included in the study medications
11. Patients unable or unwilling to comply with study protocol (e.g., alcoholism, mental illness, travel schedule)
12. Participation in a clinical study with another investigational drug in the 30 days prior to randomization or while participating in this study
13. Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2010-05-27; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert DuPont, MD, Principal Investigator — Bausch Health Americas, Inc.
Locations (12):
- Guatemala (3):
  - Santarus Investigational Site 03, Antigua Guatemala
  - Santarus Investigational Site 14, Antigua Guatemala
  - Santarus Investigational Site 04, Quetzaltenango
- Mexico (9):
  - Santarus Investigational Site 05, Guadalajara, Jalisco
  - Santarus Investigational Site 06, Cuernavaca, Morelos
  - Santarus Investigational Site 12, Cabo San Lucas
  - Santarus Investigational Site 10, Cancún
  - Santarus Investigational Site 07, Oaxaca City
  - Santarus Investigational Site 08, Puebla City
  - Santarus Investigational Site 09, Puerto Escondido
  - Santarus Investigational Site 11, Puerto Vallarta
  - Santarus Investigational Site 13, Tulum

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (two matching tablets) orally twice daily for 3 days (72 hours)
  Placebo: Placebo (two matching tablets) orally twice daily for 3 days (72 hours).
  Intent To Treat (ITT)
- Rifamycin SV MMX: Rifamycin SV MMX® 400 mg (two 200 mg tablets) orally twice daily for 3 days (72 hours).
  Rifamycin SV MMX: Rifamycin SV MMX® 400 mg (two 200 mg tablets) orally twice daily for 3 days (72 hours).
  Intent To Treat (ITT)
Period: Overall Study
Arm/Group | Placebo | Rifamycin SV MMX
Started | 65 | 199
Completed | 53 | 178
Not Completed | 12 | 21
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Use of prohibited medications | 0 | 1
Not completed — Noncompliance with study procedures | 2 | 1
Not completed — Patient required rescue medication | 8 | 17

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rifamycin SV MMX | Total
Number analyzed (Participants) | 65 | 199 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (12.72) | 28 (11.43) | 28.3 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 100 | 133
  Male | 32 | 99 | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 9 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 10 | 15
  White | 56 | 175 | 231
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Baseline Pathogen Identified [Count of Participants; unit: Participants]
  Yes | 48 | 133 | 181
  No | 17 | 66 | 83

OUTCOME MEASURES:

1. Primary Outcome: Time to Last Unformed Stool (TLUS)
Description: The primary endpoint is TLUS defined as the interval in hours between the first dose of study drug and the last unformed stool passed just before the start of Clinical Cure. An unformed stool is defined as either a soft or watery stool. TLUS will be calculated for each patient in the following manner:
  Step 1: Identify when the patient achieves Clinical Cure.
  Step 2: Moving backwards from this time, identify the time of the last unformed stool.
  Step 3: The TLUS equals the time from the first dose of study drug to the time of the last unformed stool identified in Step 2.
Time Frame: 24 hours
Population: Intent To Treat (ITT). Please note that the 75th percentile was not observed during the 120-hour study period for placebo patients.
  The percentile groups indicate the hour at which the appropriate percentage of the patient group had met the primary endpoint i.e. by 72 hours, 75% of Rifamycin SV MMX patients had met the endpoint.
Measure: Mean (95% Confidence Interval); unit: TLUS (hours)
Arm/Group | Placebo | Rifamycin SV MMX
Number analyzed (Participants) | 65 | 199
TLUS (hours)
  25th percentile | 37.4 [8.3 to 47.8] | 21. [12.7 to 25.8]
  50th percentile | 68 [48.7 to NA] — The 75th percentile was not observed during the 120-hour study period for placebo patients. | 46 [42.8 to 50.5]
  75th percentile | NA [NA to NA] — the 75th percentile was not observed during the 120-hour study period for placebo patients. | 72.2 [69 to 91.7]

2. Secondary Outcome: Clinical Cure
Description: Clinical Cure is defined as either of the following:
  * Passage of two or fewer soft stools and no watery stools, no fever (>100.4 ºF or 38 ºC), and no signs or symptoms of enteric infection (other than mild excess gas/flatulence) during a 24 hour interval in the 120-hr data collection period after the first dose of study drug
  * Passage of no stools or only formed stools and no fever during a 48-hour interval in the 120-hr data collection period after the first dose of study drug, with or without other signs or symptoms of enteric infection
Time Frame: 24 hours
Population: Intent to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rifamycin SV MMX
Number analyzed (Participants) | 65 | 199
Participants | 35 | 162

ADVERSE EVENTS:
Time Frame: The Investigator must completely and promptly record each new AE/SAE that occurs after the first dose of study drug through Visit 4 (i.e., treatment emergent AEs) on the appropriate CRF, even if the relationship of an AE to study drug is assessed by the Investigator to be "unlikely" or "not related". In addition, the investigator must document and follow SAEs that occur from Visit 4 through 30 days after the last dose of study drug.
Arm/Group | Placebo | Rifamycin SV MMX
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/199
Serious Adverse Events (participants affected / at risk) | 1/65 | 2/199
Other Adverse Events (participants affected / at risk) | 25/65 | 58/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Rifamycin SV MMX (N=199)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — investigator concluded that the event was unrelated to study medication that the neuroblastoma developed prior to enrollment in the study. No further information on outcome is available.
Abdominal pain/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Rifamycin SV MMX (N=199)
Amoebic dysentery (Infections and infestations) | 2 (2) | 0 (0)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 5 (5) | 10 (10)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 17 (17)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 10 (10)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator will provide Sponsor an opportunity of at least 30 days to review and comment on any proposed publication before it is disclosed and Sponsor shall have the right to require the removal of any Confidential Information. Sponsor shall have the right to require the publication be delayed for an additional period not to exceed 60 days to permit the filing of patent applications or to seek intellectual property protection related to information contained in such publication.